CLINICAL TRIAL: NCT01373398
Title: Phase I Clinical Trial to Evaluate the Safety and Pharmacokinetics of Intravesical Instillation of EO9 in Patients With Non-muscle Invasive Bladder Cancer(NMIBC)
Brief Title: Safety and Pharmacokinetic Study of EO9(Intravesical Instillation)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Handok Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: HD901_01
Record Dates: First submitted 2011-06-09; First posted 2011-06-15 (Estimated); Last update posted 2012-03-13 (Estimated); Status verified 2012-03

CONDITIONS: Bladder Cancer
Keywords: bladder cancer; EO9; Apaziquone
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: EO9(Apaziquone) — immediate instillation after TURBT + 6 weekly instillation 4mg/mL Apaziquone

SUMMARY:
The purpose of this study is to evaluate the safety and pharmacokinetics (PK) of intravesical instillation of EO9 in patients with non-muscle invasive bladder cancer (NMIBC).

ELIGIBILITY:
Inclusion Criteria:

* Patients who are clinically diagnosed as having stage Ta, T1, histological grade G1, G2 urothelial carcinoma of the bladder
* Patients who are confirmed to be urinary cytology negative (class I, class II) within 4 weeks prior to the present TURBT.
* P.S : 0-2 according to the ECOG.

Exclusion Criteria:

* Patients with a primary and solitary tumor.
* CIS lesions in the bladder or a history thereof.
* Grade 3 disease or a history thereof.
* Patients experiencing recurrence within 3 months following TURBT for prior NMIBC.
* Patients having stage T1 and high-grade disease.
* Invasive cancer of T2 or greater, with definite lymph node or other organ metastasis, or a history thereof.
* Patients who received intravesical chemotherapy/immunotherapy treatment within 6 months prior to the present TURBT.
* Patients who underwent systemic chemotherapy or radiotherapy whose field of exposure included the bladder.
* Patients with suspected bladder perforation at the time of the present TURBT.
* A complication of a malignant tumor of the upper urinary tract or urethra, or a history thereof.
* Malignancy within 5 years other than NMIBC (except thyroid cancer)
* A serious viral or bacterial infection within the last 4 weeks.

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2011-05; Primary Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Safety assessment based on all Adverse events(causal relationship, incidence, severity, etc.) | 14 weeks

SECONDARY OUTCOMES:
pharmacokinetics assessment of EO9 and it's metabolites in blood and urine | before, 30, 55, 90 mins of EO9 instillation

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Site 01, Seoul
  - Site 02, Seoul